CLINICAL TRIAL: NCT06306144
Title: Mild Cognitive Impairment After Minor Stroke: Evaluation of Early-phase Telecare Programs (Psychoeducation and Computerized Cognitive Stimulation)
Brief Title: Early-phase Telecare Programs for Minor Stroke
Acronym: COGaDOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL23_0691
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Minor Stroke
Keywords: cognitive complaint; computerized stimulation; psychoeducation; tele-rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients receiving the Psychoeducation Intervention (Experimental): Patients will participate in a 6-week psychoeducation telerehabilitation intervention, that will consist of two 45-minute sessions per week. Each week they will participate in a 45-minute on-line session with a rehabilitation clinician and later in the week will complete 45 minutes of exercises set by the rehabilitation clinician
  Interventions: Behavioral: Psychoeducation
- Patients receiving the Computerised Cognitive Stimulation Intervention (Experimental): Patients will participate in a 6-week cognitive stimulation telerehabilitation intervention, that will consist of two 45-minute sessions per week. Each week they will participate in a 45-minute on-line session with a rehabilitation clinician and later in the week will complete 45 minutes of on-line exercises set by the rehabilitation clinician.
  Interventions: Behavioral: Computerised Cognitive Stimulation
- Patients receiving the Usual Care (Experimental): Patients randomized to this group will complete the questionnaires and the cognitive tests but will receive no intervention
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Psychoeducation — Arm 1 : Psychoeducation aims to inform patients about post-stroke cognitive impairment, teach them coping strategies to compensate for these difficulties, provide information on symptom recognition and management, and offer emotional and psychological support to help them meet the challenges associated with these potential cognitive impairments.
  Arms: Patients receiving the Psychoeducation Intervention
Behavioral: Computerised Cognitive Stimulation — Arm 2 :Patients will participate in a 6-week cognitive stimulation telerehabilitation intervention, that will consist of two 45-minute sessions per week. Each week they will participate in a 45-minute on-line session with a rehabilitation clinician and later in the week will complete 45 minutes of on-line exercises set by the rehabilitation clinician
  Arms: Patients receiving the Computerised Cognitive Stimulation Intervention
Behavioral: Usual Care — Arm 3 : No specific care.
  Arms: Patients receiving the Usual Care

SUMMARY:
Minor strokes (few acute neurological symptoms ; NIHSS score <5), represent almost 65% of cerebrovascular ischemic events. The increasing incidence of stroke in people under 65, together with advances in diagnostic and revascularization techniques, mean that post-stroke life expectancy is now in the order of decades. Most patients with minor stroke are rapidly discharged from hospital, with follow-up focused on secondary prevention and they are offered little or no rehabilitation.

However, up to 70% of patients with minor stroke experience difficulties resuming their social or professional activities, which can lead to social and economic disruption (delayed/compromised return to work) and an increased risk of depression. While some care recommendations exist for this population, in France there is no consensus nor identified care pathway for follow-up assessment or management of these patients. Furthermore, existing services are unevenly distributed across the country, and research into the effectiveness of rehabilitation is still scarce, leading to uncertainty as to which interventions should be prioritized to decrease difficulties related to cognitive impairment.

Since there are currently no rehabilitation proposals in France for patients with mild cognitive impairment after mild stroke, in this trial the investigaror will investigate the effectiveness of two six-week telerehabilitation programs each consisting of a weekly session supervised by a therapist and a self-rehabilitation session. The aim of this multicenter randomized controlled trial is the evaluate the relevance and feasibility of early identification of patients eligible for a cognition-focused management proposal and the efficacy of two telecare programs, (a) psychoeducation and (b) computerized cognitive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, aged between 18 and 65 years old
* Hospitalization for a first stroke
* Minor stroke: NIHSS score < 5 on discharge from neurovascular unit
* Post-stroke delay < 8 weeks
* Living at home (not institutionalized)
* Affiliated with social security or benefiting from such a scheme
* French language
* Presence of a cognitive complaint (FACT-Cog "perceived cognitive impairments" subscale score < 55) and absence of major cognitive impairment
* Signature of informed consent

Exclusion Criteria:

* History of stroke
* Uncorrected hearing or visual impairment
* Neurological pathology other than stroke or disabling psychiatric disorder
* Unstabilized epilepsy
* Undergoing cognitive rehabilitation in another context or having integrated a post-stroke therapeutic education program
* Living in a white zone that does not allow for remote rehabilitation
* Unable to connect to the Internet
* Pregnant, parturient or breast-feeding women* (interview data)
* Persons deprived of their liberty by judicial or administrative decision
* Persons admitted to a health or social institution for purposes other than research
* Adults under legal protection (guardianship, curatorship)
* Taking part in other interventional research involving a period of exclusion still in progress at pre-inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to demonstrate the benefits of early management following a minor stroke on participation at 6 months post-stroke. | At the end of the study : 36 months
  Difference in the Participation score (from the Participation subscale of the stroke impact scale) between the pre-intervention evaluation and the evaluation 6 months post-stroke, between the intervention and non-intervention groups

SECONDARY OUTCOMES:
to evaluate the effects on quality of life of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs will be evaluated with quality of life measured using the WHOQOL-BREF Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.
to evaluate the effects on cognitive complaint of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs will be evaluated with cognitive complaint measured using the FACT-Cog;
  Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.
to evaluate the effects on cognitive function of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs will be evaluated with cognitive function (notably attentional, executive and memory functions) measured using a custom-designed battery of neuropsychological tests;
  Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.
to evaluate the effects on mood and anxiety of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs on mood and anxiety will be measured by the HADS
  Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.
to evaluate the effects on fatigue of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs on fatigue will be measured by the FACIT-Fatigue
  Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.
to evaluate the effects on participation of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs on participation will be measured by the score on the Participation subscale of the Stroke Impact Scale
  Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.
to evaluate the effects on health status of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs on health status will be measured by EQ-5D-5L;
  Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.
to evaluate the effects on health status of the proposed programs at post-intervention, 6 months post-stroke and 9 months post-stroke in comparison with measurements taken before the start of management (pre-intervention visit 1) | At the end of the study : 36 months
  the effects of the proposed programs on the medico-economic impact of these interventions.
  Difference in each outcome measure score between the pre-intervention evaluation and the evaluations post-intervention and at 9 months post-stroke, between the intervention and non-intervention groups.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHU Lille, Lille
  - Hôpital Henry Gabrielle, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: No